CLINICAL TRIAL: NCT07086794
Title: Targeting Immune Inflammation in Cocaine Use Disorder: A Human Laboratory Study With Pentoxifylline
Brief Title: Cocaine and Pentoxifylline (BED IN 47)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 104811; R01DA063069 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Cocaine; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will be treated daily with an oral placebo.
  Interventions: Drug: Placebo
- Pentoxifylline Dose 1 (Experimental): Subjects will be treated daily with oral pentoxifylline (1200 mg).
  Interventions: Drug: Placebo; Drug: Cocaine (IV); Drug: Pentoxifylline
- Pentoxifylline Dose 2 (Experimental): Subjects will be treated daily with oral pentoxifylline (1600 mg).
  Interventions: Drug: Placebo; Drug: Cocaine (IV); Drug: Pentoxifylline

INTERVENTIONS:
Drug: Placebo — The effects of placebo will be determined.
Drug: Cocaine (IV) — The effects of IV Cocaine will be determined.
  Arms: Pentoxifylline Dose 1; Pentoxifylline Dose 2
Drug: Pentoxifylline — The effects of pentoxifylline will be determined.
  Arms: Pentoxifylline Dose 1; Pentoxifylline Dose 2

SUMMARY:
This will be a human laboratory study evaluating the influence of pentoxifylline treatment on the effects of cocaine. Supported by and included in the Helping to End Addiction Long-term® (HEAL) Initiative.

ELIGIBILITY:
Inclusion Criteria:

1. able to speak/read English,
2. not seeking treatment for drug use at the time of the study,
3. female or male between the ages of 18 and 55 years,
4. recent smoked or intravenous cocaine use verified by benzoylecgonine positive urine, as well as fulfillment of DSM-5 diagnostic criteria for CUD,
5. judged to be medically and psychiatrically healthy by study physicians other than the diagnosis for CUD at the time of screening,
6. ECG, read by a cardiologist, within normal limits,
7. females using an effective form of birth control and not pregnant or breastfeeding and 8) no known contraindications or allergies to pentoxifylline.

Exclusion Criteria:

1. unable to speak/read English,
2. seeking treatment for drug use,
3. under 18 years or over 55 years,
4. no recent smoked or intravenous cocaine use as indicated by benzoylecgonine negative urine and no DSM-5 diagnosis of CUD,
5. judged to be medically or psychiatrically unhealthy by study physicians at the time of screening,
6. ECG, read by a cardiologist, outside normal limits,
7. females not using an effective form of birth control or pregnant or breastfeeding,
8. contraindications or allergies to pentoxifylline, and
9. Self-reported history of head trauma, seizure, CNS tumors, or use of concomitant medications that lower seizure threshold, or first-degree family history of seizures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Reinforcing Effects of Cocaine | 9 times over approximately 1 month inpatient admission
  Number of Times Subjects Choose Cocaine (Maximum of 5 Choices) Over Money

CONTACTS AND LOCATIONS:
Locations (1):
- Psychopharmacology of Addiction Laboratory, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No